CLINICAL TRIAL: NCT06917417
Title: The Effect of Laughter Therapy Given to Mothers in the Postpartum Period on Marital Adjustment, Life Satisfaction and Maternal Bonding Levels in Mothers; A Randomized Controlled Trial
Brief Title: The Effect of Laughter Therapy on Marital Adjustment, Life Satisfaction and Maternal Attachment Level in Mothers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Havva Tokgöz Kekeç, PhD Student, Msc Midwife, Selcuk University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2024/617
Record Dates: First submitted 2025-04-01; First posted 2025-04-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Postpartum; Mothers
Keywords: postpartum period; maternal attachment; life satisfaction; laughter therapy
MeSH Terms: conditions — Personal Satisfaction | interventions — Laughter Therapy

STUDY DESIGN:
Intervention Model Description: After randomisation, a WhatsApp group will be established with the mothers in the laughter therapy group. Before starting the application, the 'Zoom' programme will be downloaded to the phone or computer of the mothers in the laughter therapy group. A WhatsApp group will be formed with at least 5-10 people, and a total of 10 sessions of laughter therapy will be applied with the groups for 5 weeks, 2 sessions per week. No intervention will be made to the control group, and they will be asked to fill in the questionnaire forms simultaneously.
Who Masked: Participant, Outcomes Assessor
Masking Description: In the study, the researcher will apply the intervention to the laughter therapy group. Therefore, researcher blinding will not be performed. In the study, a single blinding method in which the participants are blinded will be used. In order to prevent detection bias, data collection forms will be collected by the interviewer who has no knowledge about the research groups. In order to prevent reporting bias, the data obtained from the research will be coded as A and B by an independent researcher and transferred to the SPSS programme, and the analysis of the data coded in terms of groups will be carried out by an independent statistical expert.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- laughter therapy group (Experimental): After randomization, a WhatsApp group will be established with the mothers in the laughter therapy group. Before starting the application, the "Zoom" program will be downloaded to the phone or computer of the mothers in the laughter therapy group. Groups will be formed with at least 5-10 people, and a total of 10 sessions of laughter therapy will be applied to the groups, 2 sessions per week for 5 weeks.
  Interventions: Behavioral: Laughter Therapy
- control group (No Intervention): The control group will not be subjected to any intervention and will be asked to fill out the questionnaire forms simultaneously.

INTERVENTIONS:
Behavioral: Laughter Therapy — A laughter yoga session; It is approximately 30 minutes and consists of four parts. These sections; hand clapping and warm-up exercises, deep breathing exercises, childish games and laughter exercises. In each laughter yoga session, the first three parts are the same, but the laughter exercises in the fourth part vary. In the first session of each new group, the introduction of laughter yoga, its purpose and objectives will be discussed. 10 minutes will be allocated for this section in the first session of each group. Therefore, the first session is planned to be 40 minutes in each group and all subsequent sessions are planned to be 30 minutes.
  Arms: laughter therapy group

SUMMARY:
The postnatal period is a fragile period with physical and psychological changes as well as hormonal changes in the mother. Mind-body based complementary practices such as yoga, meditation, relaxation exercises can be used to improve well-being and facilitate adaptation to the changes experienced during this period. Among these practices, laughter yoga is new, simple, cost-effective, non-invasive, widely available online and easily applicable/accessible. In studies, individuals in different populations from children to the elderly have proven that laughter therapy interventions cause improvement in mood and life satisfaction. Looking at the literature, studies on laughter therapy in Turkey are limited and no study has been found on this subject. Therefore, the present study aims to investigate the effect of laughter therapy given to mothers in the postnatal period on partner adjustment, life satisfaction and maternal attachment level in mothers. It is thought that this study will make a very important contribution to the literature.

DETAILED DESCRIPTION:
The postnatal period is a fragile period with physical and psychological changes as well as hormonal changes in the mother. In the transition to parenthood in the postnatal period, expectant parents experience changes that have important effects on the couple's relationship, the baby-parent relationship and the development of the baby. The positive relationship and harmony of the spouses are important in raising a child. Maternal attachment starts in the prenatal period and reaches the highest level in the postnatal period. It is known that inadequate maternal attachment to the baby poses a threat to the healthy development and well-being of the baby. Therefore, it is important to evaluate the psycho-social welfare of the mother in the postnatal period, to evaluate the level of mother-infant attachment and to make effective midwifery interventions.

Studies in the literature have documented the positive role of laughter in improving quality of life. In addition, it was determined that laughter therapy intervention during pregnancy increased the mental well-being of pregnant women and positively affected prenatal attachment levels. Laughter therapy can be used for both preventive and therapeutic purposes. Poor mental health of the mother poses a danger to the baby and the mother. Studies on laughter therapy are limited in Turkey. In order to increase evidence-based data, there is a need to investigate the potential effectiveness of laughter therapy interventions in terms of mothers' health. It is thought that this study will make a very important contribution to the literature.

ELIGIBILITY:
Inclusion Criteria:

* At least primary school graduate
* Over 18 years of age
* Volunteer to participate in the research
* Heterosexual
* With a spouse or partner
* At term
* With a single, healthy baby
* Have not had any intra-abdominal surgery
* With a 1-12 month postpartum baby
* Women who can use the Zoom program

Exclusion Criteria:

* Those who do not speak Turkish,
* Those with hearing and visual impairments,
* Those with mental disabilities,
* Those diagnosed with known psychiatric diseases,
* Mothers of babies with disabilities and chronic health problems
* Women with physical illnesses that prevent them from participating in Laughter Yoga sessions (breathing difficulties, persistent cough, vertigo, severe heart disease, hemorrhoids, any type of hernia such as neck, waist or inguinal hernia, severe back pain, urinary incontinence, epilepsy, etc.)
* Women who develop an acute health problem for themselves or their babies, who have had their mothers or babies suddenly hospitalized, who have lost their babies, who have separated from their spouses or partners, who do not attend laughter therapy sessions regularly, and who cannot be reached after the application will be excluded from the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 90 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-05-25 (Estimated); Study Completion 2025-06-25 (Estimated)

PRIMARY OUTCOMES:
Revised Dyadic Adjustment Scale | 1st Time: Day 1, 2nd Time: Day 45, 3rd Time: Day 75
  RDAS is the final 14-item form of the 32-item DAS, developed by Spanier (1976), and revised by Busby et al. (1995). Turkish validity and reliability study of the scale was conducted by Gündoğdu Psychometric evaluations of the scale in the Northern Cyprus sample were re-conducted by Bayraktaroğlu and Çakıcı. The scale was developed to assess the quality of relationships between couples who are married or in a marriage-like relationship. This questionnaire includes three subscales that are consensus (items 1, 2, 3, 4, 5, and 6), satisfaction (items 7, 9, 11, 12, and 13), and conflict (items 8, 10, and 14). The scale is 5-point Likert type and coded as 1 = Never, 2 = Rarely, 3 = Sometimes, 4 = Often, and 5 = Always. Items 7, 8, 9, and 10 of the scale are reverse scored. Scores on the RDAS range from 0 to 70 with higher scores indicating greater relationship satisfaction and lower scores indicating greater relationship distress.
Life Satisfaction Scale | 1st Time: Day 1, 2nd Time: Day 45, 3rd Time: Day 75
  It is a self-assessment scale developed by Diener et al. The scale consists of five items and is unidimensional. The scale has a Likert-type rating scale with options from 1 to 7 ranging from 'not at all appropriate' to 'very appropriate'. The scale was translated and adapted into Turkish by Köker. The highest score that can be obtained from the Life Satisfaction Scale is 35 and the lowest score is 5. A high score on the scale indicates a high degree of satisfaction and a low score indicates a low degree of satisfaction.
Maternal Attachment Inventory | 1st Time: Day 1, 2nd Time: Day 45, 3rd Time: Day 75
  Maternal Attachment ınventory was originally developed by Mary E. Muller in 1994 for the assessment of maternal attachment. The validity and reliability of the Turkish form was done by Kavlak and Şirin (2009). The scale has no sub-dimensions. Maternal attachment inventory, an indicator of and measuring affection, is a self-administered scale and can only be administered to literate women who can read and write and understand what they read. Each item is in a 4-point Likert type ranging from "always" to "never." Each item contains statements and points, showing a = 4 (always), b = 3 (often), c = 2 (sometimes), and d = 1 (never). An overall score is obtained from the sum of all items. A high score indicates a high level of maternal attachment. The lowest score to be obtained from the scale is 26, while the highest score is 104. The scale has no cutoff score. The Maternal Attachment Scale is administered to mothers who have a baby of at least 1-month old. It is not applied to pregnant wo
Personal Information Form | 1st time: Day 1
  Personal Information Form It consists of 16 questions developed by the researcher as a result of literature reviews. It consists of 11 questions about the socio-demographic characteristics of the mothers (age, education level, income status, presence of social security, etc.) and 5 questions about obstetric characteristics (number of pregnancies, parity status, etc.).

CONTACTS AND LOCATIONS:
Locations (1):
- Selçuk University Faculty of Medicine Hospital, Konya, Selçuklu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] van der Wal CN, Kok RN. Laughter-inducing therapies: Systematic review and meta-analysis. Soc Sci Med. 2019 Jul;232:473-488. doi: 10.1016/j.socscimed.2019.02.018. Epub 2019 Mar 5. PMID 31029483
- [Background] Spanier GB (1976). Measuring dyadic adjustment: A newscales for assessing the quality of marriage and similar dyads. Journal of Marriage and the Family; 38: 15-28.
- [Background] Scott JK, Nelson JA, Dix T. Interdependence among mothers, fathers, and children from early to middle childhood: Parents' sensitivity and children's externalizing behavior. Dev Psychol. 2018 Aug;54(8):1528-1541. doi: 10.1037/dev0000525. Epub 2018 Jun 21. PMID 29927264
- [Background] Quick AD, Tung I, Keenan K, Hipwell AE. Psychological Well-being across the Perinatal Period: Life Satisfaction and Flourishing in a Longitudinal Study of Black and White American Women. J Happiness Stud. 2023 Mar;24(3):1283-1301. doi: 10.1007/s10902-023-00634-6. Epub 2023 Mar 13. PMID 37273506
- [Background] Pu DF, Rodriguez CM. Spillover and Crossover Effects: Mothers' and Fathers' Intimate Partner Violence, Parent-Child Aggression Risk, and Child Behavior Problems. Child Maltreat. 2021 Nov;26(4):420-430. doi: 10.1177/1077559520985936. Epub 2021 Jan 13. PMID 33438464
- [Background] Namazinia M, Mazlum SR, Mohajer S, Lopez V. Effects of laughter yoga on health-related quality of life in cancer patients undergoing chemotherapy: a randomized clinical trial. BMC Complement Med Ther. 2023 Jun 12;23(1):192. doi: 10.1186/s12906-023-04028-2. PMID 37303065
- [Background] Muller ME. Prenatal and postnatal attachment: a modest correlation. J Obstet Gynecol Neonatal Nurs. 1996 Feb;25(2):161-6. doi: 10.1111/j.1552-6909.1996.tb02420.x. PMID 8656307
- [Background] Küçükkelepçe, DŞ, Ünver H, & Kurt N. (2024). Kahkaha Yogasının Emzirme Öz-Yeterliliği Üzerine Etkisinin İncelenmesi: Randomize Kontrollü Çalışma, Journal of Academic Research in Nursing (JAREN), 10(1).
- [Background] Kumcağız H, Aydın Avci İ, Caner Ş. (2018). Yaşam doyumu, postpartum depresyon ve özkıyım olasılığı arasındaki ilişki. Anadolu Hemşirelik ve Sağlık Bilimleri Dergisi, 21(1):1-9.
- [Background] Köker S. (1991). Normal ve Sorunlu Ergenlerin Yaşam Doyumu Düzeyinin Karşılaştırılması. Ankara Üniversitesi Sosyal Bilimler Enstitüsü. Ankara. Yayımlanmamış Yüksek Lisans Tezi.
- [Background] Ko Y, Park S. A pilot randomized controlled trial of distance laughter therapy for mothers' level of depression, anxiety, and parental stress during the COVID-19 pandemic. PLoS One. 2023 Jul 14;18(7):e0288246. doi: 10.1371/journal.pone.0288246. eCollection 2023. PMID 37450484
- [Background] Kilic S, Can R, Yilmaz SD. Spousal support and dyadic adjustment in the early postpartum period. Women Health. 2024 Feb 7;64(2):121-130. doi: 10.1080/03630242.2024.2304891. Epub 2024 Jan 30. PMID 38221674
- [Background] Kekec HT, Dikmen HA. The relationship of social support perceived by mothers and fathers and dyadic adjustment with maternal and paternal attachment in the postpartum period. Dev Psychobiol. 2023 Jan;65(1):e22358. doi: 10.1002/dev.22358. PMID 36567652
- [Background] Kavlak O, Şirin A. (2009). Maternal Bağlanma Ölçeği'nin Türk toplumuna uyarlanması. Uluslararası İnsan Bilimleri Dergisi; 6:188-202.
- [Background] Holmes EK, Sasaki T, & Hazen NL. (2013). Smooth versus rocky transitions to parenthood: Family systems in developmental context. Family Relations, 62, 824-837. 10.1111/fare.12041
- [Background] Diener E, Emmons RA, Larsen RJ, Griffin S. The Satisfaction With Life Scale. J Pers Assess. 1985 Feb;49(1):71-5. doi: 10.1207/s15327752jpa4901_13. PMID 16367493
- [Background] Dağlı, A. ve Baysal, N. (2016). Yaşam Doyumu Ölçeğinin Türkçe'ye uyarlanması: Geçerlik ve güvenirlik çalışması, Elektronik Sosyal Bilimler Dergisi, 15(59), 1250-1262.
- [Background] Si S Celi K A, Kilinc T. The effect of laughter yoga on perceived stress, burnout, and life satisfaction in nurses during the pandemic: A randomized controlled trial. Complement Ther Clin Pract. 2022 Nov;49:101637. doi: 10.1016/j.ctcp.2022.101637. Epub 2022 Jul 5. PMID 35810525
- [Background] Bayraktaroğlu HT, Çakıcı ET. (2017). Psychometric properties of Revised form Dyadic Adjustment Scale in a sample from North Cyprus. International Journal of Educational Science; 19(2,3): 113-9.
- [Background] Alves S, Fonseca A, Canavarro MC, Pereira M. Does Dyadic Coping Predict Couples' Postpartum Psychosocial Adjustment? A Dyadic Longitudinal Study. Front Psychol. 2020 Sep 25;11:561091. doi: 10.3389/fpsyg.2020.561091. eCollection 2020. PMID 33101131
- [Background] Ainsworth MDS, Blehar MC, Waters, Wall S. (2015). Patterns of Attachment Erlbaum, Hillsdale.
- [Background] Agapinar Sahin S, Bekar M. The influence of laughter yoga on pregnancy symptoms, mental well-being, and prenatal attachment: A randomized controlled study. Health Care Women Int. 2023 Jun;44(6):782-801. doi: 10.1080/07399332.2022.2164284. Epub 2023 Jan 10. PMID 36625775